CLINICAL TRIAL: NCT06164821
Title: Efficary and Safety of Luspatercept for Treatment of Anaemia in Transfusion-dependent β-thalassaemia in Southwest China
Brief Title: Clinical Observation of Luspatercept in Treatment of Chinese Adult β-thalassaemia Patients With TD β-thalassemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hematology department of the 920th hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-thal01
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Effect of Drug
Keywords: luspatercept; β-Thalassemia
MeSH Terms: interventions — luspatercept

STUDY DESIGN:
Intervention Model Description: 5 cases with transfusion burden<7.5 units/24 weeks, and 5 cases with transfusion burden 7.5-15 units/24 weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- luspatercept arm (Experimental): Luspatercept was given once subcutaneously every 3 weeks for 24 weeks in the treatment period, . Luspatercept was started at 1·0 mg/kg with titration up to 1·25 mg/kg, or reduction in the event of toxicity or excessive haemoglobin concentration increase.. During the treatment, the hemoglobin of patients before each injection of luspatercept should be monitored, and the common adverse reactions (AE) should be monitored. According to the judgment and practice of clinicians, the best supportive treatment, including blood transfusion, iron chelation therapy, and anti-infection treatment, should be provided for patients receiving luspatercept treatment. If the patient has blood transfusion, it is necessary to obtain the blood transfusion record from the hospital system.Concomitant use of iron chelating agents was also recorded.
  Interventions: Drug: luspatercept

INTERVENTIONS:
Drug: luspatercept — Adult patients with TD thalassemia were given luspatercept subcutaneous injection.

SUMMARY:
To assesse the efficacy and safety of luspatercept versus placebo in China patients with transfusion-dependent β-thalassaemia.

DETAILED DESCRIPTION:
This was a prospective, multicenter, open-label, multicenter clinical study to observe the efficacy and safety of luspatercept in the treatment of adult patients with transfusion-dependent β-thalassemia in Chinese clinical practice.

Luspatercept has been approved for listing in China for the treatment of that requires regular infusion of red blood cells and red blood cell infusion ≤ 15 units/24 weeks β- Adult patients with thalassemia. The BELIEVE study enrolled 117 patients of Asian descent from Malaysia, Thailand, Taiwan, Australia, the United States, the United Kingdom, and Canada. Efficacy results similar to those in the global intention-to-treat population were observed in Asian patients with a baseline transfusion load of 6 to 15 units per 24 weeks. The results in the Asian population provide valuable reference for the safety and efficacy of luspatercept in the Chinese population.

Ten adult patients with β-thalassemia were enrolled in this study,divided into two groups (5 cases with transfusion burden<7.5 units/24 weeks, and 5 cases with transfusion burden 7.5-15 units/24 weeks).Luspatercept was given once subcutaneously every 3 weeks for 24 weeks in the treatment period, . Luspatercept was started at 1·0 mg/kg with titration up to 1·25 mg/kg, or reduction in the event of toxicity or excessive haemoglobin concentration increase. During the treatment, the hemoglobin of the patients before each injection of luspatercept was monitored, and the common adverse reactions (AE) were monitored.The primary end point was the percentage of the LTB and HTB group patients who had a reduction in the transfusion burden of at least 33% and reduce blood transfusion unit from baseline group.According to the judgment and practice of clinicians, the best supportive treatment, including blood transfusion, iron chelation therapy, and anti-infection treatment, should be provided for patients receiving luspatercept treatment. Thus，this clinical trial is going to further explore its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old;
2. A clear diagnosis of transfusion-dependent β-thalassemia (including αβ mixed type) with red blood cell transfusion ≤15u within 24 weeks before enrollment (one unit of red blood cell in overseas clinical research is 200-350ml packed red blood cells, which should be converted according to Chinese clinical practice);
3. Voluntarily participate in the study and sign the informed consent;

Exclusion Criteria:

1. pregnant or lactating women;
2. Allergic to luspatercept and/or luspatercept for injection excipients;
3. Severe liver dysfunction: Liver enzymes (alanine aminotransferase ALT or aspartate aminotransferase AST) ≥ 3 times normal value.;
4. Severe renal injury: eGFR<30 ml/min/1.73m3 or end-stage renal disease;
5. heart disease, New York Heart Association (NYHA) class 3 or higher heart failure, or the need for treatment Severe arrhythmia, or recent myocardial infarction within 6 months;
6. The patient had uncontrolled hypertension;
7. Patients with a history of deep vein thrombosis or stroke within 24 weeks prior to enrollment.;
8. Treatment with ESA, luspatercept, thalidomide or hydroxyurea within 12 weeks before enrollment;
9. Any significant other medical condition, laboratory abnormality, or mental illness;
10. Investigators deemed enrollment inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of units in cumulative transfusion volume | Within 24 weeks
  The decrease of cumulative blood transfusion volume in low transfusion burden group (<7.5 units /24 weeks) and high transfusion burden group (7.5-15 units /24 weeks) after 24 weeks of treatment;
Proportion of patients with a 33% reduction in transfusion burden | Within 24 weeks
  33% reduction in blood transfusion burden at week 24 in low transfusion burden group (<7.5 units /24 weeks) and high transfusion burden group (7.5-15 units /24 weeks);

SECONDARY OUTCOMES:
Blood transfusion burden reduction ratio | Within 24 weeks
  The proportion of RBC transfusion burden reduced by 50% at any 12 weeks;
  (2) transfusion independence (TI) rates at any 8-week and any 12-week in the whole study population;
Ratio of TI | Within 24 weeks
  Transfusion independence (TI) rates at any 8 weeks and at any 12 weeks in the entire study population；

OTHER OUTCOMES:
Security Index | Within 33 weeks
  Vital signs, laboratory measures, adverse events (AES), and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes